CLINICAL TRIAL: NCT02514772
Title: A Randomized, Double- Blind, Controlled, Parallel-group, Multicenter Study to Assess the Safety and Immunogenicity of Transitioning to GP2013 or Re-treatment With Rituxan® or MabThera® in Patients With Active Rheumatoid Arthritis, Previously Treated With Rituxan® or MabThera®
Brief Title: GP2013 Treatment in Patients With Active Rheumatoid Arthritis, Previously Treated With Rituxan® or MabThera®
Acronym: ASSIST-RT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sandoz (Industry)
Collaborators: Hexal AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GP13-302
Record Dates: First submitted 2015-07-30; First posted 2015-08-04 (Estimated); Results first posted 2017-12-28 (Actual); Last update posted 2017-12-28 (Actual); Status verified 2017-11

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- GP2013 - proposed biosimilar rituximab (Experimental): 10 mg/mL in 500 mg (50 mL) single-use vials. For i.v. administration, two 500 mg vials (1000 mg of active molecule) of concentrate are diluted in 0.9% NaCl solution and infused i.v. The treatment course consists of 2 i.v. infusions 2 weeks apart (at Day 1 and Day 14).
  Interventions: Biological: GP2013 - A Proposed biosimilar rituximab
- Originator rituximab - Rituxan ® or MabThera ® (Active Comparator): 10 mg/mL in 500 mg (50 mL) single-use vials. For i.v. administration two 500 mg vials (1000 mg of active molecule) of concentrate are diluted in 0.9% NaCl solution and infused i.v. The treatment course consists of 2 i.v. infusions 2 weeks apart (at Day 1 and Day 14).
  Interventions: Biological: Originator rituximab - Rituxan ® or MabThera ®

INTERVENTIONS:
Biological: GP2013 - A Proposed biosimilar rituximab
  Arms: GP2013 - proposed biosimilar rituximab
Biological: Originator rituximab - Rituxan ® or MabThera ®
  Arms: Originator rituximab - Rituxan ® or MabThera ®

SUMMARY:
The study objective is to identify potential safety risks of the transition from US-licensed Rituxan® or EU-approved MabThera® to GP2013 (proposed biosimilar product) as compared to continuous treatment with the originator product in terms of general safety and immunogenicity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of rheumatoid arthritis (RA) according to ACR 2010 criteria
* Completed one full treatment course with either Rituxan® or MabThera®
* Eligible for a further treatment course with Rituxan® or MabThera®- Currently treated with methotrexate

Exclusion Criteria:

* RA functional status class IV (ACR 1991 revised criteria)
* Systemic manifestation of RA
* Positive serology for hepatitis B or hepatitis C infection
* Active systemic infection
* History of cancer
* Known severely immunocompromised state

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandoz Inc., Study Chair — Sponsor GmbH
Locations (65):
- United States (39):
  - Rheumatology Associates of North Alabama, PC, Huntsville, Alabama
  - Clinical and Translational Research Center of Alabama PC, Tuscaloosa, Alabama
  - Arizona Arthritis & Rheumatology Research, PLLC, Glendale, Arizona
  - Arizona Arthritis and Rheumatology Research, PLLC, Mesa, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Phoenix, Arizona
  - Arizona Arthritis and Rheumatology Research, PLLC, Phoenix, Arizona
  - TriWest Research Associates, LLC, El Cajon, California
  - Valerius Medical Group and Research Center of Greater Long Beach, Inc, Long Beach, California
  - Pacific Arthritis Center Medical Group, Santa Maria, California
  - Westlake Medical Research Inc., Thousand Oaks, California
  - Inland Rheumatology and Osteoporosis Medical Group, Upland, California
  - Arthritis Associates & Osteoporosis Center of Colorado Springs, Colorado Springs, Colorado
  - Denver Arthritis Clinic, Denver, Colorado
  - Bay Area Arthritis and Osteoporosis, Brandon, Florida
  - Sunrise Research Institute, Inc., Miami, Florida
  - Omega Research Consultants, LLC, Orlando, Florida
  - Arthritis Center, Palm Harbor, Florida
  - Arthritis Research of Florida, Inc., Palm Harbor, Florida
  - Southwest Florida Clinical Research Center, Tampa, Florida
  - Florida Medical Clinic, PA, Zephyrhills, Florida
  - Idaho Arthritis and Osteoporosis Clinic, Meridian, Idaho
  - Bluegrass Community Research, Inc., Lexington, Kentucky
  - Arthritis and Rheumatology Consultants, P.A., Edina, Minnesota
  - North Mississippi Medical Clinical, Inc, Tupelo, Mississippi
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - Innovative Health Research, Las Vegas, Nevada
  - Arthritis and Osteoporosis Consultants of The Carolinas, Charlotte, North Carolina
  - Physicians East, PA, Greenville, North Carolina
  - STAT Research Inc., Dayton, Ohio
  - Arthritis & Rheumatology Center of Oklahoma, PLLC, Oklahoma City, Oklahoma
  - Health Research of Oklahoma, Oklahoma City, Oklahoma
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Emkey Arthritis and Osteoporosis Clinic, PC, Wyomissing, Pennsylvania
  - Low Country Rheumatology, PA, Charleston, South Carolina
  - Piedmont Arthritis Clinic, PA, Greenville, South Carolina
  - Amarillo Center for Clinical Research, Ltd., Amarillo, Texas
  - Pioneer Research Solutions, Inc., Houston, Texas
  - Arthritis and Osteoporosis Center of South Texas, San Antonio, Texas
  - Rheumatic Disease Center, Glendale, Wisconsin
- Germany (16):
  - Praxis Prof. Herbert Kellner, München, Bavaria
  - Praxiszentrum St. Bonifatius, München, Bavaria
  - Rheumahaus - GbR, Potsdam, Brandenburg
  - Universitätsklinikum Frankfurt, Frankfurt am Main, Hesse
  - Gemeinschaftspraxis Dr. von Hinüber, Dr. Demary, Hildesheim, Lower Saxony
  - Klinikum Porz am Rhein, Cologne, North Rhine-Westphalia
  - Schwerpunktpraxis Rheumatologie, Rendsburg, Schleswig-Holstein
  - MVZ Ambulantes Rheumazentrum Erfurt, Erfurt, Thuringia
  - Rheumatology Center Prof. Neeck, Bad Doberan
  - Rheumapraxis Steglitz, Berlin
  - Immanuel Krankenhaus Berlin, Standort Berlin-Buch, Berlin
  - Rheumatologisches MVZ Dresden GmbH, Dresden
  - Rheumatologie im Struensee-Haus, Hamburg
  - LMU Klinikum der Universität München, München
  - Studienambulanz Dr. Wassenberg, Ratingen
  - Universitätsklinikum Würzburg, Würzburg
- Hungary (4):
  - Országos Reumatológiai És Fizioterápiás Intézet, Budapest
  - QUALICLINIC Kft, Budapest
  - Csongrád Megyei Dr. Bugyi István Kórház, Szentes
  - MÁV Kórház és Rendelőintézet Szolnok, Szolnok
- Poland (6):
  - Szpital Uniwersytecki Nr 2 im. Dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Twoja Przychodnia - Centrum Medyczne Nowa Sol, Nowa Sól
  - Slaskie Centrum Reumatologii, Rehabilitacji i Zapobiegania Niepelnosprawnosci im gen. Jerzego Zietka, Ustroń
  - Linea Corporis Chirurgia Plastyczna, Warsaw
  - Medycyna Kliniczna Marzena Waszczak, Warsaw
  - Centrum Medyczne AMED, Warsaw

REFERENCES:
- [Derived] Tony HP, Kruger K, Cohen SB, Schulze-Koops H, Kivitz AJ, Jeka S, Vereckei E, Cen L, Kring L, Kollins D. Brief Report: Safety and Immunogenicity of Rituximab Biosimilar GP 2013 After Switch From Reference Rituximab in Patients With Active Rheumatoid Arthritis. Arthritis Care Res (Hoboken). 2019 Jan;71(1):88-94. doi: 10.1002/acr.23771. PMID 30295429

RESULTS

PARTICIPANT FLOW:
Groups:
- GP2013: 10 mg/mL in 500 mg (50 mL) single-use vials. For i.v. administration, two 500 mg vials (1000 mg of active molecule) of concentrate are diluted in 0.9% NaCl solution and infused i.v. The treatment course consists of 2 i.v. infusions 2 weeks apart (at Day 1 and Day 14)
  GP2013 - A proposed biosimilar rituximab
  Patients in this group are switched from originator rituximab (which they received before study participation) to GP2013
- Rituxan® / MabThera®: 10 mg/mL in 500 mg (50 mL) single-use vials. For i.v. administration two 500 mg vials (1000 mg of active molecule) of concentrate are diluted in 0.9% NaCl solution and infused i.v. The treatment course consists of 2 i.v. infusions 2 weeks apart (at Day 1 and Day 14)
  Originator rituximab - Rituxan ® or MabThera ® dependent on region of participation (USA patients receive Rituxan; EU patients receive MabThera).
  Patients in this group receive same originator rituximab as they received before study participation
Period: Overall Study
Arm/Group | GP2013 | Rituxan® / MabThera®
Started | 53 | 54
Completed | 50 | 52
Not Completed | 3 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- GP2013: 10 mg/mL in 500 mg (50 mL) single-use vials. For i.v. administration, two 500 mg vials (1000 mg of active molecule) of concentrate are diluted in 0.9% NaCl solution and infused i.v.
  GP2013 - A Proposed biosimilar rituximab
- Rituxan ® / MabThera ®: 10 mg/mL in 500 mg (50 mL) single-use vials. For i.v. administration two 500 mg vials (1000 mg of active molecule) of concentrate are diluted in 0.9% NaCl solution and infused i.v.
  Originator rituximab - Rituxan ® or MabThera ® dependent on region of participation (USA patients receive Rituxan; EU patients receive MabThera)
- Total: Total of all reporting groups
Arm/Group | GP2013 | Rituxan ® / MabThera ® | Total
Number analyzed (Participants) | 53 | 54 | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 44 | 39 | 83
  >=65 years | 9 | 15 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (9.91) | 57.1 (12.14) | 57 (11.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 39 | 85
  Male | 7 | 15 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 9
  Not Hispanic or Latino | 44 | 47 | 91
  Unknown or Not Reported | 5 | 2 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 51 | 52 | 103
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 18 | 35
  Europe | 36 | 36 | 72
Weight at screening [Mean (Standard Deviation); unit: kg] | 80.12 (20.22) | 81.62 (20.46) | 80.88 (20.26)
Duration since initial diagnosis of rheumatoid arthritis [Mean (Standard Deviation); unit: years] | 13.46 (9.39) | 14.01 (8.51) | 13.74 (8.92)
C-reactive protein (CRP) at baseline [Mean (Standard Deviation); unit: mg/L] | 9.67 (24.25) | 11.64 (23.63) | 10.66 (23.84)
Dose of methotrexate at baseline [Mean (Standard Deviation); unit: mg/week] | 14.53 (6.203) | 15.46 (5.141) | 15.00 (5.684)
Prednisone equivalent steroid dose at baseline [Mean (Standard Deviation); unit: mg/day] — Population: Steroids were not taken by all patients at the study start
  mg/day
    number analyzed (Participants) | 23 | 26 | 49
    (all) | 5.39 (1.80) | 4.64 (2.36) | 4.99 (2.13)
Number of previous treatments courses with rituximab [Mean (Standard Deviation); unit: treatment course] | 4.1 (3.32) | 5.0 (3.75) | 4.6 (3.56)
Number of previous treatment courses with rituximab [Number; unit: treatment course]
  1 | 13 | 13 | 26
  >1 | 40 | 41 | 81
Experienced infusion-related reactions during rituximab treatments prior to randomization [Number; unit: participants]
  No | 51 | 51 | 102
  Yes | 2 | 3 | 5
Anti-drug antibodies (ADA) at screening [Number; unit: participants]
  Negative | 52 | 53 | 105
  Positive | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Experiencing Anaphylactic Reactions
Description: 2006 NIAID/FAAN* criteria were used for identification of anaphylactic reactions within 24h of each study drug infusion.
  For patients with no history of infusion-related reactions during their previous treatments with rituximab, symptoms/signs in at least 2 out of 4 organ systems:
  * Skin/mucosal tissue
  * Respiratory organs
  * Drop of systolic blood pressure (<90 mmHg or variance from baseline >30%) or associated symptoms
  * Gastrointestinal organs were defined as an anaphylactic reaction.
  The same criteria were also applied to patients with history of infusion-related reactions during their previous treatments with rituximab. In addition, if these patients experienced only a rapid drop in systolic blood pressure (<90 mmHg or variance from baseline >30%), this was defined as an anaphylactic reaction disregarding involvement of other organ systems.
  * NIAID - National Institute of Allergy and Infectious Diseases FAAN - Food Allergy and Anaphylaxis Network
Time Frame: Within 24 hours of each study drug infusion: on Day 1 and Day 14
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Groups:
- GP2013: 10 mg/mL in 500 mg (50 mL) single-use vials. For i.v. administration, two 500 mg vials (1000 mg of active molecule) of concentrate are diluted in 0.9% NaCl solution and infused i.v.
  GP2013 - A proposed biosimilar rituximab
  Patients in this group are switched from originator rituximab (which they received before study participation) to GP2013
- Rituxan® / MabThera®: 10 mg/mL in 500 mg (50 mL) single-use vials. For i.v. administration two 500 mg vials (1000 mg of active molecule) of concentrate are diluted in 0.9% NaCl solution and infused i.v.
  Originator rituximab - Rituxan ® or MabThera ® dependent on region of participation (USA patients receive Rituxan; EU patients receive MabThera).
  Patients in this group receive same originator rituximab as they received before study participation
Arm/Group | GP2013 | Rituxan® / MabThera®
Number analyzed (Participants) | 53 | 54
Participants | 0 | 1
Statistical Analysis 1: Comparison: GP2013 vs Rituxan® / MabThera®; Test type: Other; Difference (%) = -1.9, 95% CI 2-sided [-20.6 to 16.9]

2. Primary Outcome: Number of Patients Experiencing Hypersensitivity Reactions
Description: The standardized MedDRA query (SMQ) - Hypersensitivity reactions (SMQ 20000214) was used for the identification of hypersensitivity reactions overall from first infusion in the adverse event database.
Time Frame: 24 weeks study duration
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | GP2013 | Rituxan® / MabThera®
Number analyzed (Participants) | 53 | 54
Participants | 5 | 6
Statistical Analysis 1: Comparison: GP2013 vs Rituxan® / MabThera®; Test type: Other; Difference (%) = -1.7, 95% CI 2-sided [-20.6 to 16.9]

3. Primary Outcome: Immunogenicity
Description: Number of patients tested positive for anti-drug-antibodies (ADA) post-randomization.
  Patients with negative ADA results at screening and at least one evaluable post-randomization ADA assessment are included in the analysis
Time Frame: 24 weeks study duration
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | GP2013 | Rituxan® / MabThera®
Number analyzed (Participants) | 51 | 53
Participants | 0 | 1
Statistical Analysis 1: Comparison: GP2013 vs Rituxan® / MabThera®; Test type: Other; Difference (%) = -1.9, 95% CI 2-sided [-21.2 to 17.6]

4. Primary Outcome: Number of Patients Experiencing Potential Infusion-Related Reactions
Description: Patients, experienced infusion related reactions repeatedly (i.e. during the first and second infusion) are counted only once in the overall line.
Time Frame: On the day of and on the day after each study drug infusion (e.g. on study day 1 and 2 for the 1st study drug infusion and on study day 14 and 15 for the 2nd study drug infusion, if the second drug infusion was given on study day 14)
Population: The total number of patients, who received second infusion in GP2013 arm differs from the total number of patients in GP2013 arm due to patients withdrawn after the 1st infusion.
Measure: Count of Participants; unit: Participants
Arm/Group | GP2013 | Rituxan ® / MabThera ®
Number analyzed (Participants) | 53 | 54
Participants
  On day of or on day after first infusion | 4 | 7
  On day of or on day after second infusion: number analyzed (Participants) | 51 | 54
  On day of or on day after second infusion | 2 | 5
  Overall on day(s) of or after either infusion | 6 | 10
Statistical Analysis 1: Comparison: GP2013 vs Rituxan ® / MabThera ®; Incidence difference of infusion-related reactions, occurred on day of or on day after first infusion (i.e. on study day 1 or on study day 2); Test type: Other; Mean Difference (Final Values) = -5.4, 95% CI 2-sided [-24.2 to 13.3]
Statistical Analysis 2: Comparison: GP2013 vs Rituxan ® / MabThera ®; Incidence difference of infusion-related reactions, occurred on day of or on day after second infusion (i.e. on study day 14 or on study day 15); Test type: Other; Mean Difference (Final Values) = -5.3, 95% CI 2-sided [-24.5 to 13.6]
Statistical Analysis 3: Comparison: GP2013 vs Rituxan ® / MabThera ®; Incidence difference of infusion-related reactions overall on day(s) of or day(s) after either infusion (i.e. on day 1 or 2 and on day 14 or day 15); Test type: Other; Mean Difference (Final Values) = -7.2, 95% CI 2-sided [-26.0 to 11.4]

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) are reported from Day 1 until the end of study (Week 24)
Arm/Group | GP2013 | Rituxan® / MabThera®
All-Cause Mortality (participants affected / at risk) | 0/53 | 1/54
Serious Adverse Events (participants affected / at risk) | 0/53 | 3/54
Other Adverse Events (participants affected / at risk) | 19/53 | 21/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GP2013 (N=53) | Rituxan® / MabThera® (N=54)
Atrial fibrillation (Cardiac disorders) | 0 | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 0 | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 (1)
Fibrin D dimer increased (Investigations) | 0 | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GP2013 (N=53) | Rituxan® / MabThera® (N=54)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 3 (3)
Bronchitis (Infections and infestations) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (4)
Nasopharyngitis (Infections and infestations) | 2 (3) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Headache (Nervous system disorders) | 2 (3) | 2 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor shall have the right to the first publication or presentation of the results of the study which is intended to be a joint, multi-center publication of the study results. Following the first publication, institutions and/or Principal Investigators may publish or present data or results from the study per the terms of the clinical trial agreement.